CLINICAL TRIAL: NCT05288465
Title: Hair Repigmentation in Patients Undergoing on Cerebrolysin Treatment for Neurological Diseases.
Brief Title: Hair Repigmentation During Cerebrolysin Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Collaborators: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Roberto Montes de Oca Luna, Principal Investigator, Universidad Autonoma de Nuevo Leon
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NC15-001
Record Dates: First submitted 2022-02-16; First posted 2022-03-21 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Hair Problems
Keywords: Hair graying
MeSH Terms: conditions — Hair Diseases | interventions — cerebrolysin

STUDY DESIGN:
Intervention Model Description: Longitudinal study of hair repigmentation in patients receiving cererbolisin treatment for neurological diseases
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hair repigmentation during Cerebrolysin treatment for neurological diseases (Experimental): Patients prescribed for Cerebrolysin treatment due neurological diseases.
  Interventions: Drug: Cerebrolysin

INTERVENTIONS:
Drug: Cerebrolysin — Patients prescribed for Cerebrolysin treatment due neurological disease are invited to donate a scalp punch biopsy prior to and after completing the prescribed treatment.
  Other Names: Renacenz

SUMMARY:
Open-label histological study of scalp biopsies from patients undergoing treatment with Cerebrolysin as therapy for cerebrovascular disease. The aim is to assess by histological techniques the causes of follicular repigmentation that occurs during the Cerebrolysin treatment.

DETAILED DESCRIPTION:
Patients who fulfill the study requirements will receive the standard Cerebrolysin protocol as follows: Intravenous (iv) infusions of 5 vials per week, 2 vials on Mondays and 3 vials on Thursdays for 4 weeks, followed by an 8-week resting period prior to the next cycle of treatment. Each patient will receive 3 cycles giving a total of 9 months of follow-up. For intravenous infusions, each 10 ml vial containing 215.2mg / ml of Cerebrolysin (Ever Pharma) is diluted with physiological saline solution (NaCI 0.9%) to a final volume of 100 mL.

A pre- and post-treatment biopsies will be collected from the achromotrichia area of each patient. Antisepsis of the area will be performed prior to each biopsy with chlorhexidine, followed by local anesthesia with lidocaine 2% and epinephrine. The biopsy will be collected using a 4mm punch and the wound will be sutured with non-absorbable stitches with Prolene 4-0.

ELIGIBILITY:
Inclusion Criteria:

* Known neurologist prescription for Cerebrolysin treatment due ischemic or hemorrhagic stroke, traumatic brain injury or dementia.
* Age-related white or gray hair.
* Above 40 years old
* Voluntarily consents in written informed consent by the principal or legal representative

Exclusion Criteria:

* Patients with a diagnosis of Chronic Kidney Disease (CKD).
* Known history of seizures, epilepsy, or hypersensitivity to one or any drug components.
* Pregnant patients.
* Patients with a history of recent treatment of hair coloring products.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-06-02 (Actual); Primary Completion 2015-12-07 (Actual); Study Completion 2016-12-23 (Actual)

PRIMARY OUTCOMES:
Macroscopic evaluation of scalp repigmentation | From the beginning of the treatment until 9th month.
  Change in scalp pigmentation throughout cerebrolysin treatment measured by gray/white hair score.
Microscopic evaluation of scalp repigmentation | From the beginning of the treatment until 9th month.
  Change in melanin production in the scalp measured by histochemical staining score.
Evaluation of scalp melanocytes function. | From the beginning of the treatment until 9th month.
  Change in melanocyte function activity measured by immunostaining score.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario. Dr. José Eleuterio González, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No